CLINICAL TRIAL: NCT06977867
Title: The Effect of Stress Ball Use on Comfort, Anxiety, and Patient Satisfaction in Hemodialysis Patients
Acronym: Stress Ball
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Hasret Topalı, Lecturer, Bitlis Eren University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/8-2 and E.6610
Record Dates: First submitted 2025-04-24; First posted 2025-05-18 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Hemodialysis Patients
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress Ball (Experimental): All hemodialysis patients who meet the inclusion criteria will be asked to squeeze a stress ball during their dialysis sessions (3 times a week for 1 month, totaling 12 sessions). Anxiety, comfort, and patient satisfaction levels will be assessed using three measurements: a pre-test before the intervention, a mid-test at the end of the 6th session (2nd week), and a post-test after the 12th session. Patients will be instructed to use the stress ball throughout their dialysis session. They will be asked to squeeze the ball for at least 10-15 minutes during each session.
  Interventions: Device: Stress Ball
- Control (Other): The hemodialysis patients in the control group will not use the stress ball and will receive standard care throughout the study period. Similar to the intervention group, levels of anxiety, comfort, and patient satisfaction will be assessed at three time points: prior to the intervention (pre-test), at the end of the second week (after the 6th session), and at the end of the fourth week (post-test, after the 12th session).
  Interventions: Other: standard care

INTERVENTIONS:
Device: Stress Ball — All hemodialysis patients who meet the inclusion criteria will be asked to squeeze a stress ball during their dialysis sessions (3 times a week for 1 month, totaling 12 sessions). Anxiety, comfort, and patient satisfaction levels will be assessed using three measurements: a pre-test before the intervention, a mid-test at the end of the 6th session (2nd week), and a post-test after the 12th session. Patients will be instructed to use the stress ball throughout their dialysis session. They will be asked to squeeze the ball for at least 10-15 minutes during each session.
  Arms: Stress Ball
Other: standard care — The hemodialysis patients in the control group will not use the stress ball and will receive standard care throughout the study period. Similar to the intervention group, levels of anxiety, comfort, and patient satisfaction will be assessed at three time points: prior to the intervention (pre-test), at the end of the second week (after the 6th session), and at the end of the fourth week (post-test, after the 12th session).
  Arms: Control

SUMMARY:
Chronic kidney disease represents a significant public health issue both in Türkiye and worldwide, with the majority of patients undergoing hemodialysis treatment. Individuals receiving hemodialysis often experience not only physical discomfort but also psychological distress, including heightened anxiety and reduced comfort. The aim of this study is to evaluate the effects of stress ball use on comfort, anxiety, and patient satisfaction among hemodialysis patients. The stress ball is a simple and cost-effective non-pharmacological intervention that aids individuals in managing stress by redirecting their attention. Notably, this study is unique in simultaneously investigating comfort, anxiety, and satisfaction parameters within this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Being literate
* Having no visual or hearing impairments
* Being able to communicate verbally
* Having no physical disability that would prevent the use of a stress ball
* Not having a diagnosed anxiety disorder and not using medication for it
* Willingness to participate in the study

Exclusion Criteria:

* Currently using sedative medications
* Having a diagnosed psychiatric disorder
* Having any physical limitation that prevents squeezing a stress ball

Ages: 18 Years to 98 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Level of anxiety | 1 month
  The anxiety levels of patients included in the study will be assessed prior to the intervention using the Visual Analog Scale (VAS). The VAS scores will be categorized as follows: low anxiety (0-3), moderate anxiety (4-6), and high anxiety (7-10).
Patient's comfort | 1 month
  The comfort levels of patients using the stress ball during the hemodialysis procedure will be assessed using the Hemodialysis Comfort Scale. The minimum score obtainable from the scale (20) indicates low comfort, while the maximum score (100) reflects high comfort.
Level of patient satisfaction | 1 month
  Patient satisfaction during the hemodialysis procedure among those using the stress ball will be assessed using the Visual Analog Patient Satisfaction Scale. VAS scores will be categorized as follows: low satisfaction (0-3), moderate satisfaction (4-6), and high satisfaction (7-10).

CONTACTS AND LOCATIONS:
Locations (1):
- Bitlis State Hospital, Bitlis, Tatvan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liyanage T, Ninomiya T, Jha V, Neal B, Patrice HM, Okpechi I, Zhao MH, Lv J, Garg AX, Knight J, Rodgers A, Gallagher M, Kotwal S, Cass A, Perkovic V. Worldwide access to treatment for end-stage kidney disease: a systematic review. Lancet. 2015 May 16;385(9981):1975-82. doi: 10.1016/S0140-6736(14)61601-9. Epub 2015 Mar 13. PMID 25777665